CLINICAL TRIAL: NCT03409120
Title: Unlocking Dystonia From Parkinson's Disease With Directional DBS Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Harrison Walker, MD, Associate Professor of Neurology, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-300001136
Record Dates: First submitted 2018-01-13; First posted 2018-01-24 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-07

CONDITIONS: Dystonia-Parkinsonism, Adult-Onset; Parkinson Disease
Keywords: Dystonia; Parkinson's Disease
MeSH Terms: conditions — Dystonia-Parkinsonism, Adult-Onset; Parkinson Disease; Dystonia

STUDY DESIGN:
Intervention Model Description: To measure the effects of directional DBS on dystonia, we will measure the change in the Burke-Fahn-Marsden Dystonia Rating Scale at 2, 4, 6, and 12 months after surgery versus preoperative baseline
Masking Description: This study will run in conjunction with "Biomarkers to Guide Directional DBS for Parkinson's Disease" (ClinicalTrials.gov Identifier: NCT03353688). It is a double blinded study investigating the effectiveness of directional DBS leads in which participants and some investigators will have no knowledge of the DBS settings participants experience.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Dystonia Severity Assessment (Experimental): We will measure the effects of DBS on dystonia by assessing changes in the Burke-Fahn-Marsden Dystonia Rating Scale at 2, 4, 6, and 12 months after surgery to implant the Boston Scientific Vercise PC IPG with directional DBS lead versus preoperative baseline.
  Interventions: Device: Boston Scientific Vercise PC IPG with directional DBS lead

INTERVENTIONS:
Device: Boston Scientific Vercise PC IPG with directional DBS lead — We will contrast the effects of omnidirectional versus directional STN DBS on dystonia symptoms in patients with PD.

SUMMARY:
This study occurs during five visits that are already scheduled as part of "Biomarkers to Guide Directional DBS for Parkinson's Disease" (ClinicalTrials.gov Identifier: NCT03353688). If participants have dystonia associated with Parkinson's disease, the investigators will consent and administer one additional rating scale (Burke-Fahn-Marsden Dystonia Rating Scale) to assess the severity of dystonia.

DETAILED DESCRIPTION:
To measure the effects of DBS on dystonia, the investigators will measure the change in the Burke-Fahn-Marsden Dystonia Rating Scale at 2, 4, 6, and 12 months after surgery versus preoperative baseline. This will allow them to contrast the effects of omnidirectional versus directional STN DBS on dystonia symptoms in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in "Biomarkers to Guide Directional DBS for Parkinson's Disease" (ClinicalTrials.gov Identifier: NCT03353688)
* Diagnosis of Parkinson's disease with and without dystonia

Exclusion Criteria:

* Not enrolled in "Biomarkers to Guide Directional DBS for Parkinson's Disease" (ClinicalTrials.gov Identifier: NCT03353688)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harrison C Walker, MD, Principal Investigator — Associate Professor of Neurology
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Olson JW, Nakhmani A, Irwin ZT, Edwards LJ, Gonzalez CL, Wade MH, Black SD, Awad MZ, Kuhman DJ, Hurt CP, Guthrie BL, Walker HC. Cortical and Subthalamic Nucleus Spectral Changes During Limb Movements in Parkinson's Disease Patients with and Without Dystonia. Mov Disord. 2022 Aug;37(8):1683-1692. doi: 10.1002/mds.29057. Epub 2022 Jun 14. PMID 35702056

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and studied prospectively as part of the SUNDIAL (SUbthalamic Nucleus DIrectionAL stimulation) study, a randomized, double-blind crossover study contrasting directional versus circular unilateral STN DBS for PD (FDA Investigational Device Exemption G-170063). Further details on inclusion/exclusion are outlined at https://clinicaltrials.gov/ct2/show/NCT03353688.
Pre-assignment Details: All subjects provided written informed consent prior to participation with approval from the institutional review board. We included data from all consecutively enrolled participants. Dystonia status was not part of the enrollment criteria.
Period: Overall Study
Arm/Group | Dystonia Severity Assessment
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Patients Enrolled in Study: All patients enrolled in the study
Arm/Group | Study Patients Enrolled in Study
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Burke-Fahn-Marsden Total Dystonia Scale [Mean (Standard Deviation); unit: units on a scale] | 3.5 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Burke-Fahn-Marsden Dystonia Rating Scale
Description: Evaluation of degree of dystonia related symptoms. Domains evaluated include eyes, mouth, speech/swallowing, neck, arms, trunk, and legs. Each domain is scored on degree of provoking factor (0= no dystonia at rest or with action; 4 = dystonia present at rest) and severity factor (0 = no dystonia; 4 = extreme/severe dystonia). Scores are then weighted yielding a total score between 0 and 120. Higher scores on the scale indicate greater disease severity.
Time Frame: 5 minutes
Population: We analyzed data from all enrolled participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Patients Enrolled in Study
Number analyzed (Participants) | 38
units on a scale | 3.5 (6.0)
Statistical Analysis 1: Comparison: Study Patients Enrolled in Study; We tested the equivalence of Burke-Fahn-Marsden scores over time (at baseline and at two time periods following DBS surgery) using a repeated measures ANOVA; Test type: Superiority; p < 0.001, linear mixed effects model

ADVERSE EVENTS:
Time Frame: 1 year from baseline visit
Arm/Group | Dystonia Severity Assessment
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

LIMITATIONS AND CAVEATS:
Time and physical constraints during surgery sometimes limit data collection, and acute implant of the DBS lead introduces microlesion effects that could alter electrophysiology.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT03409120/Prot_000.pdf
  • Informed Consent Form (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT03409120/ICF_001.pdf